CLINICAL TRIAL: NCT00679887
Title: Chronic Shoulder Pain of Myofascial Origin,a Randomised Clinical Trial Using Ischemic Compression Therapy.
Brief Title: Chronic Shoulder Pain Treated by Pressures With the Thumbs on the Trigger Points
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guy Hains Chiropractor (Other)
Responsible Party: Guy Hains chiropractor, UQTR
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CER-05-102-07.05
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Shoulder Pain
Keywords: chiropractic; myofascial trigger points; ischemic compression; shoulder pain
MeSH Terms: conditions — Shoulder Pain | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Ischemic compression on trigger points located around the shoulder. Active comparator. Ischemic compression, 5 weeks
  Interventions: Procedure: ischemic compression

INTERVENTIONS:
Procedure: ischemic compression — Active Comparator, ischemic compression, 3 times a week,5 weeks

SUMMARY:
The purpose of this study is to find the efficacy of treating the trigger points located around the shoulder in patients suffering from chronic shoulder pain.

DETAILED DESCRIPTION:
Chronic shoulder pain is a common condition which should be treated by surgery only wen conservative approaches have been tried. in the present trial the authors intend to find the effectiveness of treating the triggers points located in muscles, ligaments and tendons surrounding the shoulderin patients suffering from chronic shoulder pain.

The technique used in this trial is ischemic compression(thumb tip pressure) on the trigger points

ELIGIBILITY:
Inclusion Criteria:

* 30 to 60 years old.
* To have suffered from shoulder pain on a daly basis for at least 3 months
* Participants had to be able to raise the arm above ther head.
* They had accept to receive 15 chiropractic treatments without charge.

Exclusion Criteria:

* Past surgery to the arm.
* Injection to the shoulder in the month preceding the trial.
* A diagnosis of rheumatoid arthritis or any other systemic disorders affecting the joints.
* Shoulder pain from an herniated disc.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2003-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index questionnaire | At baseline, after 15 treatments ,30 days aftr the treatments and 6 months later

SECONDARY OUTCOMES:
Pain visual analog scale | After 15 treatments, 30 days after the treatments and 6 months later.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Hains, DC, Principal Investigator — UQTR; Martin Descarreaux, DC, PHD, Study Chair — UQTR
Locations (1):
- 2930 Cote Richelieu, Trois-Rivières, Quebec, Canada